CLINICAL TRIAL: NCT02485197
Title: A Pilot Study Investigating Differences in Muscle Metabolic Function in Individuals Aged 65-75 Years With Different Vitamin D Status Before and After 7-days of Aerobic Training
Brief Title: Muscle Metabolic Function in Older Adults With Different Vitamin D Status Before and After Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Travis Thomas (Other)
Responsible Party: Sponsor-Investigator, David Travis Thomas, Ph.D., RD, CSSD, CSCS, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 12-1029-F6A
Record Dates: First submitted 2013-04-25; First posted 2015-06-30 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Vitamin D Deficiency
Keywords: Muscle Metabolic Function; Vitamin D Status; 25(OH)D; Older Adults
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low 25(OH)D (Other): We will recruit individuals with low 25(OH)D (<30ng/mL).
  Interventions: Other: 7 continuous days of aerobic training
- High 25(OH)D (Other): We will recruit individuals with higher 25(OH)D (at least 20ng/mL units higher then that of the "low 25(OH)D group).
  Interventions: Other: 7 continuous days of aerobic training

INTERVENTIONS:
Other: 7 continuous days of aerobic training — For 7 consecutive days, subjects will perform up to 45 minutes of exercise consisting of treadmill walking at a progressive intensity of about 60-65% of their maximum heart rate. This heart rate range is estimated to be below 60% VO2 max.

SUMMARY:
This is a small pilot aerobic training trial designed to examine differences between normal-high and low vitamin D levels and 7-days of aerobic training on local VO2 measured by non-invasive Hybrid Diffuse Optical Spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* 65-75 years of age

Exclusion Criteria:

* Currently have or have a history of cardiovascular or pulmonary disease that would preclude the involvement in the performance of exercise.
* Uncontrolled diabetes or hypertension.
* History of neurological conditions related to spinal derangement, disk disease, peripheral neuropathies, tremor and rigidity
* History of leg/hip trauma, inflammation, infection rhabdomyolysis, or leg surgery in the past 3 months
* Have a diagnosis of osteoporosis (as determined by DXA)
* Participated in a resistance or aerobic training program in the last 3 months
* Engage in more than 1 hr/week of vigorous activity
* Body mass index >29
* On hormone replacement therapy

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Muscle VO2 consumption | Up to 3 months
  The objective is to examine the difference in gastrocnemius VO2 consumption in individuals that either have normal-high or low 25(OH)D and are undergoing 7-days of a treadmill training program.

CONTACTS AND LOCATIONS:
Overall Officials: David T Thomas, PhD, Principal Investigator — University of Kentucky; Maja Redzic, MS, Study Director — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States